CLINICAL TRIAL: NCT06429878
Title: The Long Term Effect of MRI Before Radical Prostatectomy.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Erik Rud, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 248365
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: disease-free survival; overall survival; functional outcomes
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were randomized to either MRI or no-MRI before radical prostactomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no-MRI (Active Comparator): received no MRI before prostatectomy
  Interventions: Diagnostic Test: Biparametric prostatic MRI
- MRI (Experimental): received MRI before prostatectomy
  Interventions: Diagnostic Test: Biparametric prostatic MRI

INTERVENTIONS:
Diagnostic Test: Biparametric prostatic MRI

SUMMARY:
A randomized clinical trial conducted by Oslo University Hospital between 2010 and 2012 included 438 patients with prostate cancer to the non-MRI group (216) or the MRI group (222) before robot-assisted radical prostatectomy (RALP). The primary endpoint was to compare the nerve-sparing surgery types and the proportion of positive surgical margins (PSM) in each group. The MRI group underwent more non-nerve sparing surgery, whereas the proportion of PSM was similar in both groups (p=0.4) [1]. Since the long-term effects of preoperative MRI are unknown, we aimed to assess the variations in the long-term functional and oncological outcomes between the groups.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the oncological and functional outcomes in a 12-year follow-up after RALP in patients preoperatively randomized to no-MRI or MRI.

Material: a total of 438 consecutive patients were referred to RALP. Of these, 222 were randomized to preoperative MRI (intervention group), and 216 were randomized to no MRI (control group). All underwent radical prostatectomy between 2010 and 2012.

Study design: An experimental interventional study with 12-years follow-up

Endpoints: PSA recurrence (PSA ≥0.2ng/ml) Predictors for PSA recurrence (PSM, DÁmico risk group, Gleason score, T-stage) Overall survival (OS) Predictors for OS (PSM, DÁmico risk group, Gleason score, T-stage) MRI predictors for PSM, PSA recurrence and OS

Erectile function (IEEF-5) and urinary continence (IPSS-10) Urinary incontinence rates (≥1daily pads)

Statistics: Before RALP, included patients were randomized to the i) non-MRI group and ii) MRI-group. Kaplan Meier curves express the RFS and OS in the two groups, and the Log-rank test assesses any difference. Cox regression analyses is used to calculate the effect of MRI (Hazard ratios with 95% CIs). Chi-square test is used to assess the difference in incontinence rates, and the Mann-Whitney U test for assessing the difference in median IIEF-5 and IPSS-10 scores. Binary and Cox regression analysis is used to assess the predictive value of a positive surgical margin on PSA recurrence, and the effect of MRI variables in predicting RFS and OS (ADC, tumor volume, and radiological T-classification).

Data collection and handling of data: All patients were included in the study "Clinical impact of MRI in patients with prostate cancer." The urological and/or oncological clinic have followed these patients as part of routine clinical practice. Relevant clinical data are recorded in the "Radical prostatectomy registry ." All patients have already answered appropriate questionnaires during their regular follow-up.

PhD project: The study is a PhD project for radiologist Daniyal Noor at Oslo University Hospital

ELIGIBILITY:
Inclusion Criteria:

Prostate cancer scheduled for prostatectomy. All participated in the previous RCT

Exclusion Criteria:

Patients who did not sign the consent paper for any reason or did not accept the study premises.

Patients who underwent MRI prior to randomization. Patents who withdrew their consent for any reason during the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 12-years after surgery
  The difference between patients randomized to MRI or no-MRI

SECONDARY OUTCOMES:
Overall survival (OS) | 12-years after surgery
  The difference between patients randomized to MRI or no-MRI
Erectile dysfunction | After 12 years
  The difference between patients randomized to MRI or no-MRI
The impact of the length of positive surgical margin and Gleason score upon DFS. | After 12 years
  Predictors for recurrence
The impact of MRI variables for predicting PSM, PSA recurrence and OS | After 12 years
  MRI predictors for recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rud, MD,PhD, Principal Investigator — Oslo University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rud E, Baco E, Klotz D, Rennesund K, Svindland A, Berge V, Lundeby E, Wessel N, Hoff JR, Berg RE, Diep L, Eggesbo HB, Eri LM. Does preoperative magnetic resonance imaging reduce the rate of positive surgical margins at radical prostatectomy in a randomised clinical trial? Eur Urol. 2015 Sep;68(3):487-96. doi: 10.1016/j.eururo.2015.02.039. Epub 2015 Mar 23. PMID 25813692
- See also: A link to the original study — http://clinicaltrials.gov/study/NCT01347320